CLINICAL TRIAL: NCT04607395
Title: Pre-operative Radiograph of Deep Carious Lesions as a Predictive Tool for Pulpal Exposure.
Acronym: R2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: R2_2020
Record Dates: First submitted 2020-07-23; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-07

CONDITIONS: Deep Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pre-operative radiographs of deep carious lesion
  Interventions: Radiation: pre-operative radiograph

INTERVENTIONS:
Radiation: pre-operative radiograph — Three hundred and sixty pre-operative radiographs of deep carious lesions and a "contrasted" version of the same set have been screened and annotated by 4 evaluators. Annotations were placed at the dentino-enamel junction, at the floor of the carious lesions, and on pulp chamber wall. From these annotations, the ratios residual dentin thickness/ total dentin thickness were derived. First, inter-evaluator agreement and concordance were assessed. A logistic regression that accounted for measurement error was applied to precisely estimate the capacity of the ratio to predict exposure (reported as odds-ratio).

SUMMARY:
Preserving pulpal vitality is a major challenge when excavating deep caries lesions without severe symptomatology. Pulpal exposure alters success of the treatment (dropping from 93% for indirect pulp treatment with selective excavation to 11% for direct pulpotomy) and thus prognosis of dental organ and cost-effectiveness of the treatment. The preoperative x-ray is a complementary examination which allows to estimate the depth of the carious lesion. In clinical practice, it is currently difficult to accurately measure this depth on preoperative radiographs. This lack of precision leads to a decrease in the effective capacity of the operator to predict the risk of pulpal exposure. Their interpretation is considered imprecise and is not used as a diagnostic element.

The aim of this study was to determine if the use of pre-operative retroalveolar radiographs can help to predict pulpal exposure risk.

ELIGIBILITY:
Inclusion Criteria:

-pre-operative radiographs of deep carious lesions treated with DECAT protocole, unless they were out of the study.

Exclusion Criteria:

* Impossibility to assess carious lesion on radiograph, and amalgam restorations that impairs correct examination of carious lesion
* Radiographs of poor quality and screen captures

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pre-operative radiographs of deep carious lesions treated with DECAT
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of residual dentin thickness and total dentin thickness on standard pre-operative radiographs | Outcome measure was assessed trough study completion, an average of 1 year.
  The radiographic assessment consisted in determining the depth of each carious lesion from the pre-operative radiographs and from their contrasted version. In this work, the depth of one carious lesion was measured by the ratio (expressed in percent): 100*residual dentin thickness (RDT)/ Total dentin thickness (TDT). A logistic regression that accounted for measurement error was applied to precisely estimate the capacity of the ratio to predict exposure (reported as odds-ratio).

CONTACTS AND LOCATIONS:
Locations (1):
- Professeur des Universités- Praticien Hospitalier, Lyon, France

REFERENCES:
- [Derived] Gasqui MA, Perard M, Decup F, Monsarrat P, Turpin YL, Villat C, Gueyffier F, Maucort-Boulch D, Roche L, Grosgogeat B. Place of a new radiological index in predicting pulp exposure before intervention for deep carious lesions. Oral Radiol. 2022 Jan;38(1):89-98. doi: 10.1007/s11282-021-00530-w. Epub 2021 May 5. PMID 33954908